CLINICAL TRIAL: NCT06391827
Title: A Double-blind, Placebo-controlled, Randomized, Phase 1 Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Orally Administered DA-7503 After Single and Multiple Ascending Dose Regimens in Healthy Adult and Elderly Participants
Brief Title: A Study to Evaluate Safety, Tolerability, and PK of DA-7503 in Healthy Adult and Elderly Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA7503_AD_Ia
Record Dates: First submitted 2024-04-21; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- [Single dose] DA-7503 (Experimental): 6 subjects in each Cohort(Cohort 1-5)
  Interventions: Drug: DA-7503 Single dose
- [Single dose] Placebo (Placebo Comparator): 2 subjects in each Cohort(Cohort 1-5)
  Interventions: Drug: Placebo Single dose
- [Multiple dose] DA-7503 (Experimental): 6 subjects in each Cohort(Cohort 1-4)
  Interventions: Drug: DA-7503 Multiple dose
- [Multiple dose] Placebo (Placebo Comparator): 2 subjects in each Cohort(Cohort 1-4)
  Interventions: Drug: Placebo Multiple dose

INTERVENTIONS:
Drug: DA-7503 Single dose — Oral administration for once; Dose strength is different for each cohort(Cohort 1, 2, 3, 4 and 5).
  Arms: [Single dose] DA-7503
Drug: DA-7503 Multiple dose — Oral administration once daily for 7 days; Dose strength or target volunteer is different for each cohort(Cohort 1,2,3, and 4)
  Arms: [Multiple dose] DA-7503
Drug: Placebo Single dose — Oral administraion for once.
  Arms: [Single dose] Placebo
Drug: Placebo Multiple dose — Oral administration once daily for 7 days
  Arms: [Multiple dose] Placebo

SUMMARY:
This is a double-blind, placebo-controlled, randomized, phase 1 study to evaluate safety, tolerability, and pharmacokinetics of orally administered DA-7503 after single and multiple ascending dose regimens in healthy adult and elderly participants

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers(Age: 19~55 years, 65~85 years)
2. Body weight≥50.0kg, 18.0kg/m²≤BMI≤30.0kg/m²

Exclusion Criteria:

1. Clinically significant Medical History
2. Allergy or Drug hypersensitivity
3. AST, ALT, Total billurbin > Upper Normal Range*1.5, eGFR<60mL/min/1.73m²
4. Positive for serum test results(hepatitis B, hepatitis C, HIV, syphilis test)
5. Heavy smoker(more than 10 cigarettes/day)
6. Heavy caffeine intake(more than 5 units/day)
7. Heavy alcohol intake(more than 210g/week)

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-05-07 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics of DA-7503 single dose oral administration | 5 days
  Peak Plasma Concentration of DA-7503 (Cmax)
Pharmacokinetics of DA-7503 single dose oral administration | 5 days
  Area under the plasma concentration versus time curve of DA-7503 (AUClast)
Pharmacokinetics of DA-7503 multiple dose oral administration | 11 days
  Peak Plasma Concentration of DA-7503 (Cmax)
Pharmacokinetics of DA-7503 multiple dose oral administration | 11 days
  Area under the plasma concentration versus time curve of tau (AUCtau)
Pharmacokinetics of DA-7503 multiple dose oral administration | 11 days
  Peak Plasma Concentration of DA-7503 in steady state (Cmax,ss)
Pharmacokinetics of DA-7503 multiple dose oral administration | 11 days
  Area under the plasma concentration versus time curve of tau in steady state (AUCtau,ss)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea